CLINICAL TRIAL: NCT01367314
Title: A Phase IIa, Double Blind, Randomized, Sequential Group Study to Evaluate the Safety and Efficacy of Topical NVC-422 Dermal Gel in Impetigo
Brief Title: Safety and Efficacy of Topical NVC-422 Gel in Impetigo
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: NovaBay Pharmaceuticals, Inc. (Industry)
Collaborators: Novum Pharmaceutical Research Services (Industry); International Dermatology Research, Inc. (Other)
Responsible Party: Kenneth D. Krantz, MD, PhD, NovaBay Pharmaceuticals, Inc
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CL0901
Record Dates: First submitted 2011-06-03; First posted 2011-06-07 (Estimated); Last update posted 2011-06-07 (Estimated); Status verified 2011-06

CONDITIONS: Impetigo
MeSH Terms: conditions — Impetigo | interventions — NVC-422

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- NVC-422 Dermal Gel, 1.5% (Experimental)
  Interventions: Drug: NVC-422
- NVC-422 Dermal Gel, 0.5% (Experimental)
  Interventions: Drug: NVC-422
- NVC-422 Dermal Gel, 0.1% (Experimental)
  Interventions: Drug: NVC-422

INTERVENTIONS:
Drug: NVC-422 — Dermal Gel applied 3 times per day for 7 days
  Other Names: Sodium salt of 2-(dichloroamino)-2-methylpropane-1-sulfonate monohydrate

SUMMARY:
This is a randomized, double-blind study comparing 0.1% NVC-422, 0.5% NVC-422 and 1.5% NVC-422 topical gel in children with impetigo.

DETAILED DESCRIPTION:
This study is a randomized, sequential group, double-blind study. The first 60 subjects enrolled will be randomized to either 0.1% NVC-422 or 0.5% NVC-422. Randomization is 1:2 where 20 subjects will receive 0.1% NVC-422 and 40 subjects will receive 0.5% NVC-422. If there are no safety issues regarding the first 2 doses tested, the next 60 subjects will be randomized to either 0.1% or 1.5% NVC-422 with 20 subjects receiving 0.1% and 40 subjects receiving 1.5% NVC-422.

The lesion most representative of the subject's infection will be identified as the target lesion. This target lesion will be photographed, graded clinically, and its location recorded. At Visit 1, Screening and/or Baseline, a Gram stain will be performed to assess presence of Gram-positive cocci. If Gram-positive cocci are present, a swab for culture and sensitivity will be obtained. Treatment will began immediately after randomization.

Treatment will be 3 times per day (TID) for 7 consecutive days, following a morning, afternoon, and evening schedule.

After the start of treatment (Day 1), subjects will be assessed for safety on Day 4 (± 1). Clinical and bacteriological assessments of the target lesion will also occur on Day 8 (+1) and Follow-up on Day 15 (± 2).

ELIGIBILITY:
Inclusion Criteria:

* Subjects must be 2 - 12 years of age
* Parents or Legal Guardians must sign a written informed consent document
* Positive Gram stain of target lesion showing Gram-positive cocci;
* Clinical diagnosis of primary non-bullous impetigo as per the protocol
* Skin Infection Rating Scale total score of at least 4, with at least three of the five primary signs and symptoms present at baseline including a score of 1 or greater for exudate/pus;
* Screening within one day of enrollment into the study.

Exclusion Criteria:

* Presence of other skin diseases at or near the investigational target area to be treated;
* Disease is so widespread or severe that, in the opinion of the investigator, oral antibiotic treatment is needed
* Active impetigo lesions greater than 5 cm2
* Signs and symptoms of a current infection requiring antibiotic treatment
* Use of systemic or topical antibiotics or steroids within 72 hours prior to study entry
* Females of childbearing potential

Ages: 2 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 129 (Actual)
Dates: Start 2009-08; Primary Completion 2010-05 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Clinical Response | End of Treatment (Day 8) and Follow-up (Day 15)
  Sufficient resolution of signs and symptoms of infection of the target lesion such that no additional antimicrobial therapy is required to treat the impetigo as evidenced by the SIRS score of 0 each for exudate/pus, crusting and pain and 0 or 1 each for erythema/inflammation and itching for a clinical success or a SIRS score of 0 for exudate/pus but does not meet all the criteria for clinical success for a clinical improvement.

SECONDARY OUTCOMES:
Bacteriological Response | End of Treatment (Day 8) and Follow-up (Day 15)
  The causative pathogen isolated from the target lesion at Baseline (Staphylococcus aureus and/or Streptococcus pyogenes) are eliminated on culture, or response is such that no material was available for culture and therefore is evidence of pathogen eradication.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth D. Krantz, MD, PhD, Study Director — NovaBay Pharmaceuticals, Inc.; Daisy M. Blanco, MD, Principal Investigator — Instituto Dermatológico; Jesús Feris-Iglesias, MD, Principal Investigator — Hospital Infantil Dr. Robert Reid Cabral
Locations (2):
- Dominican Republic (2):
  - Hospital Infantil Dr. Robert Reid Cabral, Santo Domingo
  - Instituto Dermatológico, Santo Domingo